CLINICAL TRIAL: NCT03805503
Title: Determination of the Minimum Local Anesthetic Dose (MLAD) of Spinal Chloroprocaine for Inguinal Herniorrhaphy in Ambulatory Surgery
Brief Title: Chloroprocaine for Inguinal Herniorrhaphy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Hospital, Ghent (Other)
Responsible Party: Sponsor
Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: EC/2014/1264
Record Dates: First submitted 2018-12-04; First posted 2019-01-15 (Actual); Last update posted 2019-01-15 (Actual); Status verified 2019-01

CONDITIONS: Spinal Anesthesia
Keywords: Chloroprocaine; spinal anesthesia; one-day clinic
MeSH Terms: interventions — chloroprocaine

STUDY DESIGN:
Intervention Model Description: Prospective, up-down sequential allocation
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- chloroprocaine 1% injectable solution (Experimental): Prospective, up-down sequential allocation : first patient receives 50mg intrathecal chloroprocaine 1%.
  An effective result will decrease the test dose of chloroprocaine with 2 mg for the next patient in this study.
  An ineffective result will increase the test dose of chloroprocaine with 2 mg for the next patient in this study.
  Interventions: Drug: Chloroprocaine 1% Injectable Solution

INTERVENTIONS:
Drug: Chloroprocaine 1% Injectable Solution — standard CSE procedure in outpatients for inguinal hernia. The first spinal dose of chloroprocaine 1% to start with is 50mg. This dose has been successfully used for spinal anesthesia in hernia repair outpatients to reach an adequate analgesia. 2,5 microgram of sufentanil will be added for prolongation of the analgesia. The testing interval is 2 mg.
  Efficacy of the analgesia will be evaluated:
  Successful : sensory block at or above T6 dermatome bilateral at the beginning of surgery without additional analgesia during surgery. Unsuccessful: sensory block under T6 dermatome bilateral and/or VAPS is more than 10 mm at the beginning of surgery what necessitates additional epidurals analgesia.
  Patients who indicate an ineffective result will receive a rescue treatment by the administration of 5 ml chloroprocaine 3% epidural every 5 minutes with maximum of 30ml. When CSE fails, general anesthesia will be performed.
  Other Names: chloroprocaine 3%

SUMMARY:
This study is to determine the minimum effective dose for intrathecal chloroprocaine in inguinal herniorrhaphy in outpatients using a Combined Spinal Epidural (CSE) anesthesia.

DETAILED DESCRIPTION:
A standard CSE procedure will be conducted in which the patient is placed in an upright sitting position on the side of the operation table and a epidural Tuohy needle 18G will be inserted into L3-L4 interspace via a loss-of-resistance technique. The dura will be punctured using a 27-gauge pencil-point spinal needle and a certain dose of chloroprocaine 1% will be given. After the spinal needle is withdrawn, an epidural catheter will be placed and the epidural needle will be withdrawn. After fixation of catheter the patient will be placed in a supine position.

The first spinal dose of chloroprocaine 1% to start with is 50mg. This dose has been successfully used for spinal anesthesia in hernia repair outpatients to reach an adequate analgesia. Each time there will be added 2,5 microgram of sufentanil for prolongation of the analgesia. The testing interval is 2 mg.

ELIGIBILITY:
Inclusion Criteria:

* Outpatients for unilateral inguinal hernia repair
* ASA I - II - III

Exclusion Criteria:

* hypersensitivity to amino-ester local anesthetics, para-aminobenzoic acid or sufentanil
* contraindications to spinal or epidural anesthesia
* bilateral inguinal herniorrhaphy
* extremes of height and weight (BMI 20 or 35 kg/m2, height 150 cm or 185 cm)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2015-09-16 (Actual); Primary Completion 2017-09-07 (Actual); Study Completion 2018-12-04 (Actual)

PRIMARY OUTCOMES:
The dose of chloroprocaine 1% needed for the individual patient for a sensory anesthesia block at or above the T6 dermatome | start of surgery
  MLAD of chloroprocaine 1% with 2,5 mcg of sufentanil needed for the individual patient required for a sensory anesthesia at or above the T6 dermatome at the beginning of surgery with no additional epidural anesthesia required during surgery

SECONDARY OUTCOMES:
Peak block height | during surgery
  highest sensible block
Time for regression of two segments | during surgery
  Time for regression of two segments
Ambulation time | From starting hour of spinal anesthesia to hour of first ambulation after the end of surgery measured up to 6 hours after surgery
  motor recovery
Time to micturition | From starting hour of spinal anesthesia to hour of first micturition after the end of surgery measured up to 6 hours after surgery
  Time to micturition
Incidence of side effects (perioperative hypotension, respiratory depression, neurologic deficits) | perioperative
  Incidence of side effects (perioperative hypotension, respiratory depression, neurologic deficits)
Time to discharge | From starting hour of spinal anesthesia to hour of discharge from hospital measured up to 6 hours after surgery
  Time to discharge
Patient satisfaction with anesthesia method: questionnaire | postoperatively,at moment of hospital discharge measured up to 6 hours after surgery
  Patient satisfaction with simple questionnair (highly satisfied, satisfied, unsatisfied)

CONTACTS AND LOCATIONS:
Overall Officials: Aliaksandra Parashchanka, MD, Principal Investigator — stafmember department of Anesthesiology

IPD SHARING:
Plan to Share IPD: No